CLINICAL TRIAL: NCT05514288
Title: Endoscopic Weight Loss Therapy: Clinical Outcomes Over One Year of Follow-up
Brief Title: Benefits of Endoscopic Bariatric Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Kenneth Park, MD, Assistant Professor of Medicine Cedars-Sinai Medical Center, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002145
Record Dates: First submitted 2022-08-18; First posted 2022-08-24 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic sleeve gastroplasty/Transoral outlet reduction (Other)
  Interventions: Procedure: Endobariatric procedure

INTERVENTIONS:
Procedure: Endobariatric procedure — Endoscopic sleeve gastroplasty or transoral outlet reduction

SUMMARY:
This 12-months long pilot study will include patients undergoing an endoscopic procedure (endoscopic sleeve gastroplasty [ESG] or transoral outlet reduction [TORe]) as clinically indicated, and subsequent follow up clinic visits for up to one year.

DETAILED DESCRIPTION:
The purpose the research is to better understand the effects of endoscopic bariatric therapy (EBT) on the weight change, hormonal changes and changes in the quality of life parameters for patients undergoing endoscopic bariatric procedures.

The primary research procedures are:

* EBT procedure (endoscopic sleeve gastroplasty [ESG] or transoral outlet reduction [TORe])
* Behavioral intervention consisting of diet therapy, exercise therapy, and behavior modification
* Collection of blood to evaluate changes in hormonal profiles

ELIGIBILITY:
Inclusion Criteria:

* Patients who are considering undergoing EBT for weight loss
* Patients with a BMI >30 kg/m2 (without obesity related comorbidities)
* Patients with a BMI >27 kg/m2 (with obesity related comorbidities)
* Patients willing and able to comply with study requirements for follow-up
* Patients who previously underwent bariatric surgery who failed to lose the expected weight or regained weight
* Individuals 18 years old or older are included

Exclusion Criteria:

* Pre-existing esophageal stenosis/stricture preventing advancement of an endoscope during screening/baseline Esophagogastroduodenoscopy (EGD)
* Esophageal, gastric or duodenal malignancy
* Severe medical comorbidities precluding endoscopy, or limiting life expectancy to less than 2 years in the judgment of the endoscopist
* Uncontrolled coagulopathy or inability to be off anticoagulation or anti-platelet medication (ASA, Plavix) for 1 week prior to and 2 weeks after each endoscopy
* Known portal hypertension, visible esophageal or gastric varices, or history of esophageal varices
* General poor health, multiple co-morbidities placing the patient at risk, or otherwise unsuitable for trial participation at the discretion of the investigator
* Pregnant or planning to become pregnant during period of study participation
* Patient refuses or is unable to provide written informed consent
* Prior surgical or endoscopic anti-reflux procedure
* Patients who are unwilling or unable to comply with the follow-up study schedule

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Changes in body weight after various endoscopic bariatric therapies | Baseline/pre-procedure, 1 month, 3 months, 6 months, and 1 year post procedure
  The investigators will compare mean percentage total body weight loss to baseline, at 1 month, 3 months, 6 months and 1 year post procedure.

SECONDARY OUTCOMES:
Changes in hormonal profiles after various endoscopic bariatric therapies | Baseline/pre-procedure, 3 months, 6 months
  Repeated blood draws will be performed, and the following hormones will be measured: ghrelin, glucagon-like peptide 1 (GLP-1), peptide YY (PYY), gastric inhibitory polypeptide (GIP), and oxyntomodulin. We will compare changes over time in hormonal levels after EBT to baseline, 3 months, and 6 months post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Park, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Liliana Bancila, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No